CLINICAL TRIAL: NCT04694638
Title: The Use of Combined Prone Positioning and High-Flow Nasal Cannula, and Non-invasive Positive Pressure Ventilation to Prevent Intubation in Acute Hypoxemic and/or Hypercapnic Respiratory Failure Secondary to COVID-19 Infection: A Feasibility, Safety Phase One, Open Label Study
Brief Title: Use of Combined Prone Positioning and High-Flow Nasal Cannula, and Non-invasive Positive Pressure Ventilation to Prevent Intubation in COVID-19 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gustavo A. Cortes Puentes, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-003191
Record Dates: First submitted 2020-07-14; First posted 2021-01-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Prone Positioning; Covid19; Hypoxemic Respiratory Failure; ARDS; Non Invasive Ventilation; High Flow Nasal Cannulla
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HFNC and NIPPV (Experimental): Combined use of prone positioning and non-invasive positive pressure ventilation (NIPPV) and high-flow nasal cannula (HFNC)
  Interventions: Other: Body position change

INTERVENTIONS:
Other: Body position change — combined use of prone positioning and high-flow nasal cannula (HFNC) and non-invasive positive pressure ventilation (NIPPV) can reduce the rate of intubation in acute hypoxemic and/or hypercapnic respiratory failure secondary to COVID-19 infection.

SUMMARY:
This research aims to understand if prone positioning combined with high-flow nasal cannula (HFNC) or non-invasive positive pressure ventilation (NIPPV) safely reduce the rate of intubation in acute hypoxemic and/or hypercapnic respiratory failure secondary to COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed COVID19 infection or suspected COVID19 infection.
* Patients requiring HFNC or NIPPV
* Patients who are clinically stable and able to tolerate the changes in position that are routinely conducted as part of the standard of care in the medical ICU.
* Patient should be able to provide informed consent to the study. Any participant speaking any language will be offered participation.
* Able to actively participate in Assisted Manual Pronation Therapy per nursing assessment.

Exclusion Criteria:

Contraindication for prone positioning:

* Intracranial pressure >30 mm Hg or cerebral perfusion pressure <60 mmHg
* Massive hemoptysis requiring an immediate surgical or interventional radiology procedure
* Tracheal surgery or sternotomy during the previous 15 days
* Serious facial trauma or facial surgery during the previous 15 days
* Deep venous thrombosis treated for less than 2 days
* Cardiac pacemaker inserted in the last 2 days
* Unstable spine, femur, or pelvic fractures
* Hemodynamic instability or severe cardiac arrhythmia (chronic AFib is not a contraindication). Mean arterial pressure lower than 60 mm Hg, >1 vasopressor agent or Norepinephrine equivalent dose >0.06 mcg/kg/min
* Pregnant women
* Single anterior chest tube with air leaks
* Burns on more than 20 % of the body surface
* Delirium or altered mental status increasing fall risk while in prone position.
* End-of-life decision before inclusion
* Subject deprived of freedom, minor, subject under a legal protective measure
* Unable to actively participate in Assisted Manual Pronation Therapy per nursing assessment
* Lacking capacity to provide informed consent.
* Individuals with mechanical or vascular disease precluding safe displacement of the head, for example: cervical spinal fusion, limited range of motion, or severe vascular occlusive disease of the head and neck.
* Body mass index (BMI) greater than 70 kg/m2, or unable to actively participate in Assisted Manual Pronation Therapy per nursing assessment at any BMI value.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Rate of intubation | 1 year
  Number of critically ill patients with acute hypoxemic and/or hypercapnic respiratory failure, secondary to COVID-19 infection to require intubation and mechanical ventilation

SECONDARY OUTCOMES:
Incidence of hypotension and cardiac arrhythmias and other nursing-related risks of combining prone positioning with high-flow nasal cannula and non-invasive positive pressure ventilation | 1 year
  To evaluate the the incidence of hypotension and cardiac arrhythmias and other nursing-related risks of combining prone positioning with high-flow nasal cannula and non-invasive positive pressure ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Cortes Puentes, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials